CLINICAL TRIAL: NCT01269957
Title: Halitosis and Mouth Breathing in Children
Status: Completed | Type: Observational
Sponsor: University of Nove de Julho (Other)
Responsible Party: Lara Jansiski Motta, Nove de Julho University
Other Study IDs: HMB029/2009
Record Dates: First submitted 2011-01-03; First posted 2011-01-04 (Estimated); Last update posted 2011-01-04 (Estimated); Status verified 2010-08

CONDITIONS: Mouth Breathing; Halitosis
Keywords: halitosis; pediatric dentistry; mouth breathing
MeSH Terms: conditions — Mouth Breathing; Halitosis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Mouth breathing
- Nasal breathing

SUMMARY:
Objective: determine whether there is a correlation between halitosis and mouth breathing in children. Study design: Fifty-five children between three and 14 years of age were divided into two groups (nasal and mouth breathing) for the assessment of halitosis. Descriptive analysis was carried out regarding the degree of halitosis in each group. The chi-square test was used for the comparison between groups, with 5% level of significance.

ELIGIBILITY:
Inclusion Criteria:

All children registered at the clinic of the specialization course in pediatric dentistry of the ABCD/SP in 2008 were included in the study.

Exclusion Criteria:

-

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All children registered at the clinic of the specialization course in pediatric dentistry of the ABCD/SP in 2008 were included in the study.
  The children were divided into two groups based on breathing pattern (nasal and mouth) for the evaluation of halitosis. Breathing pattern was determined by a clinical evaluation and specific tests (mirror test and water-in-mouth test) and confirmed by the evaluation of an otolaryngologist.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lara Motta, Principal Investigator — Nove de Julho University
Locations (1):
- Nove de Julho University, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Motta LJ, Bachiega JC, Guedes CC, Laranja LT, Bussadori SK. Association between halitosis and mouth breathing in children. Clinics (Sao Paulo). 2011;66(6):939-42. doi: 10.1590/s1807-59322011000600003. PMID 21808855